CLINICAL TRIAL: NCT02811705
Title: Life Quality Study for PFAPA Patient
Acronym: PFAPA
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Véronique Hentgen, Dr, Versailles Hospital
Other Study IDs: P15/13_PFAPA
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: PFAPA Syndrome
MeSH Terms: conditions — Marshall syndrome | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PFAPA group: Life quality for PFAPA patient report by themselves or parent
  Interventions: Other: Quality of life
- FMF group: Life quality for FMF patient report by themselves or parent
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — Quality of life

SUMMARY:
This cohort study aims to assess the quality of life (or welfare) related to the health of children and adolescents with an non genetics auto-inflammatory disease PFAPA or Marshall syndrome to compare it to children or adolescents with recurrent fever genetics of Familial Mediterranean fever (FMF) in order to improve their overall care.

ELIGIBILITY:
Inclusion Criteria:

* PFAPA syndrome patients or FMF patients

Exclusion Criteria:

* Participation refusal

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with PFAPA syndrome compare to patient with FMF syndrome
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Compare quality of life from patients with PFAPA and FMF, reported by parents and by patients themselves | 1 day

SECONDARY OUTCOMES:
Evaluate the fatigue status of patients through questionnaire PedsQL TM 3.0 multidimensional scale tiredness | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre hospitalier de Versailles, Le Chesnay
  - CH de Bicètre, Paris